CLINICAL TRIAL: NCT04042233
Title: Intraosseous Vancomycin in Primary Total Hip Arthroplasty - Designing a Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Terry Clyburn, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00022651
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prosthetic Joint Infection; Vancomycin; Joint Diseases
Keywords: total hip arthroplasty; vancomycin; intraosseous vancomycin
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV administration of vancomycin (Active Comparator): Standard IV vancomycin administration protocol.
  Interventions: Drug: Standard IV administration of vancomycin
- IO Vancomycin 500mg in 250 mL NS (Experimental): Experimental Intraosseous administration protocol.
  Interventions: Drug: Experimental Intraosseous vancomycin 500mg in 250 mL NS

INTERVENTIONS:
Drug: Experimental Intraosseous vancomycin 500mg in 250 mL NS — 500mg of Vancomycin in 250 mL of normal saline will be injected into a pre-specified region of the greater trochanter during primary total hip arthroplasty.
  Arms: IO Vancomycin 500mg in 250 mL NS
Drug: Standard IV administration of vancomycin — IV antibiotics (cefepime & vancomycin) are started in pre-op approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg, generally 1000-1750mg in 500 mL NS).
  Arms: IV administration of vancomycin

SUMMARY:
The objective of this study is to evaluate a novel vancomycin intraosseous administration protocol vs a standard IV vancomycin administration protocol for primary total hip arthroplasty patients.

DETAILED DESCRIPTION:
Patients are randomized to one of two groups.

GROUP A - Will receive IV antibiotics (cefepime & vancomycin) are started in pre-op approximately 1 hour prior to incision vancomycin dose weight-based at approximately 15mg/kg, generally 1000-1750mg in 500 milliliters (mL) normal saline (NS).

GROUP B - Will have IV cefepime started in pre-op within 1 hour of incision. Intraosseous (IO) administration of vancomycin (500mg in 250 milliliters NS) will be administered in the OR after sterile prep and draping has occurred. Injection will take place into the greater trochanter (within a pre-specified region).

Both Groups will be monitored during surgery and immediately post-operatively for adverse injection reactions (i.e. Red Man Syndrome). Both groups will otherwise follow identical post-operative protocols (including post-operative antibiotic administration).

TISSUE SAMPLES Five (5) tissue samples will be taken from each patient, 2 soft tissue samples and 3 bone samples will be taken throughout the course of the procedure.

One blood sample will be taken in both groups intraoperatively at the time of initiation of closure.

These samples will immediately be sent to a lab for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing a primary total hip arthroplasty
* Patient gives informed consent to participate in the study.
* Age Range >18

Exclusion Criteria:

* Previous surgery on the hip (including hip scopes)
* BMI above 35
* Contraindication to receiving vancomycin or cefepime (allergy, medical issue, etc)
* Inability to locate the greater trochanter or administer the IO infusion
* Refusal to participate
* Diabetes
* Immunocompromised or immunosuppressed patients (HIV, Hep C, End stage renal disease, dialysis, transplant, chemo/radiation treatment in last 6 months, medications).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry A Clyburn, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Administration of Vancomycin | IO Vancomycin 500mg in 250 mL NS
Started | 11 | 12
Completed | 10 | 10
Not Completed | 1 | 2
Not completed — 1st sample used for calibration of vancomycin tissue/bone concentration | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Administration of Vancomycin | IO Vancomycin 500mg in 250 mL NS | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.51 (5.99) | 67.89 (4.10) | 68.31 (4.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
The American Society of Anesthesiologists (ASA) physical status classification [Mean (Standard Deviation); unit: units on a scale] — ASA I A person in good health. ASA II A mild but well-managed or treated condition ASA III A serious condition that has an impact on a person's overall health. ASA IV A severe condition that's life-threatening. ASA V A life-threatening condition that needs immediate surgery to increase survival odds.
  ASA VI A deceased person who is an organ donor.
  units on a scale | 2.6 (0.52) | 2.4 (0.52) | 2.5 (0.51)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.36 (4.68) | 27.85 (4.88) | 27.6 (4.66)

OUTCOME MEASURES:

1. Primary Outcome: Systemic Vancomycin Level - Start of Case
Description: vancomycin blood level before the time of incision - typically taken approximately 10 minutes before incision.
Time Frame: approximately 10 minutes before incision
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- IV Group: IV group
- IO Group: IO
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
ug/mL | 27.98 (13.67) | 0 (0)

2. Primary Outcome: Systemic Vancomycin Level - End of Case
Time Frame: end of surgical case
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
ug/mL | 21 (7.34) | 5.75 (2.86)

3. Primary Outcome: Vancomycin Concentration of Pulvinar Soft Tissue
Description: vancomycin concentration (ug/mL) of pulvinar soft tissue. Vancomycin tissue concentration measured by high performance liquid chromotagraphy.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 7 | 7
ug/mL | 61.58 (46.64) | 71.79 (48.15)

4. Primary Outcome: Vancomycin Concentration of Intramedullary Bone
Description: Vancomycin Concentration of Intramedullary Bone in units ug/mL. Vancomycin tissue concentration measured by high performance liquid chromotagraphy.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
ug/mL | 33.93 (26.86) | 59.39 (28.43)

5. Secondary Outcome: Soft Tissue Vancomycin Level - Start of Case
Description: at start , soft tissue. Vancomycin tissue concentration (ug/mL) measured by high performance liquid chromatography.
Time Frame: at start of case within 15 minutes after incision
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
ug/mL | 63.77 (33.70) | 69.08 (37.48)

6. Secondary Outcome: Femur Vancomycin Concentration Level
Description: Intraoperative femur bone sample measured for vancomycin concentration (ug/mL). Vancomycin tissue concentration measured by high performance liquid chromatography.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
ug/mL | 20.90 (20.81) | 41.45 (29.92)

7. Secondary Outcome: Acetabulum Vancomycin Level
Description: Intra-operative Acetabulum bone vancomycin concentrations (ug/mL) measured by high performance liquid chromatography.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
ug/mL | 67.97 (24.82) | 130.88 (45.40)

8. Secondary Outcome: 30-Day Complications
Description: Complications 30 days post surgery eg. infection.
Time Frame: From the administration of antibiotics perioperatively to 30 days post op.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
Participants | 3 | 0

9. Secondary Outcome: 90-Day Complications
Description: Complications 90 days post surgery eg. infection
Time Frame: From the administration of antibiotics perioperatively to 90 days post op.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

10. Secondary Outcome: Soft Tissue Vancomycin Level - End of Case
Description: soft tissue taken at end of case, right before wound closure is initiated. Vancomycin tissue concentration (ug/mL) measured by high performance liquid chromatography.
Time Frame: right before wound closure is initiated at the end of the case
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IV Group | IO Group
Number analyzed (Participants) | 10 | 10
ug/mL | 57.14 (29.49) | 78.22 (26.25)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | IV Group | IO Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Group (N=10) | IO Group (N=10)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — 17 days post-op patient fell off some steps outside their home. Fall was mechanical in nature. Patient unable to weight bear afterwards. XR showed Vancouver B2 fracture. Patient underwent revision THA. After careful review, deemed unrelated AE.
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient went to ED for rectal bleeding.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Group (N=10) | IO Group (N=10)
serosanguinous drainag (Musculoskeletal and connective tissue disorders) | 1 (8) | 0 (0) — Patient had small part of distal incision with serosanguinous drainage 8 days post-op. By day 16 day post-op) the incision had stopped draining w/ no overlying erythema etc at any point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT04042233/Prot_001.pdf